CLINICAL TRIAL: NCT00177047
Title: Autologous Transplantation for Multiple Myeloma
Brief Title: Autologous Transplant for Multiple Myeloma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004LS001; MT2003-13 (Other: Blood and Marrow Transplantation Program); 0312M54569 (Other: IRB, University of Minnesota); NCT00293306 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Multiple Myeloma
Keywords: stem cell transplantation; chemotherapy; multiple myeloma; autologous
MeSH Terms: conditions — Multiple Myeloma | interventions — Stem Cell Transplantation; Bone Marrow Transplantation; Cyclophosphamide; Mesna; Melphalan; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy and Transplant Treatment (Experimental): Patients receiving peripheral blood stem cell mobilization, chemotherapy (cyclophosphamide + Mesna, growth factor (Granulocyte-colony stimulating factor) and autologous Peripheral Blood Stem Cell transplant with high dose melphalan (200 mg/m^2). Post-transplant maintenance therapy is then prescribed if appropriate.
  Interventions: Procedure: Stem Cell Transplant; Drug: Cyclophosphamide + Mesna; Drug: Melphalan; Biological: Granulocyte-colony stimulating factor

INTERVENTIONS:
Procedure: Stem Cell Transplant — As part of the stem cell transplant process, patients receive high doses of chemotherapy and/or radiation to treat their underlying disease, such as cancer. As one of its effects, this treatment also kills the healthy stem cells that are already in the marrow. The transplant provides new stem cells for the patient from a healthy donor; that replace the bone marrow and allow the blood counts to recover.
  Other Names: Bone Marrow Transplant
Drug: Cyclophosphamide + Mesna — Cyclophosphamide: 4mg/m^2 + Mesna. Mesna is used to reduce the undesired side effects of certain chemotherapy drugs.
  Other Names: Cytoxan
Drug: Melphalan — Administered intravenously 200 mg/m^2
  Other Names: Alkeran
Biological: Granulocyte-colony stimulating factor — Administered intravenously 10 ug/kg/day pretransplant then 5 ug/kg/day post-transplant.
  Other Names: G-CSF

SUMMARY:
This is a study of a regimen of melphalan and autologous stem cells for patients with multiple myeloma. We hypothesize that this particular regimen will improve the survival of these patients.

DETAILED DESCRIPTION:
Before starting treatment in this study, the bone marrow transplant (BMT) doctor will check the subject's general health. Subjects will have the following tests and evaluations to find out if they can participate:--Medical history and physical examination, including height and weight.--Blood tests (approximately 4 - 5 tablespoons) --Urine tests--Chest x-ray--Electrocardiogram (ECG or EKG)--Heart Scan (MUGA)--Pulmonary Function Test (PFT)--Bone marrow biopsies and aspirates. --If Female subjects of child-bearing age will have a serum pregnancy test performed. After eligible patients have been completely staged and exercised consent, they may undergo one cycle of chemotherapy (cyclophosphamide and Mesna) and growth factor (G-CSF) to effect cytoreduction and mobilization of PBSC for collection. All patients will receive high-dose melphalan followed by an autologous stem cell transplant (SCT). Blood tests will be performed frequently to evaluate the subject's response to treatment and possible side effects of treatment. If necessary, platelet and red cell transfusions will be given to maintain adequate levels and antibiotics will be given to treat or prevent infection. Subjects may also require intravenous nutritional support and pain medications during or after transplantation. The study coordinators will collect health information over three years. They will collect information every week for 100 days, then at 6 months, 1 year, 2 years, and 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the Durie and Salmon criteria for initial diagnosis of multiple myeloma, requiring therapy and meeting one of the following:

  * After initial therapy in either first complete or partial remission or no objective response
  * After achieving initial response and later disease progression, patient will be eligible after subsequent therapy upon achievement of either complete or partial response
* Is not eligible or has refused any protocols of higher priority
* 18 - 75 years of age
* Adequate organ function defined as:

  * Hematologic: hemoglobin ≥ 8 gm/dl (untransfused), white blood cells (WBC) ≥ 3000/μl, absolute neutrophil count (ANC) ≥ 1500/μl, platelets ≥ 100,000/μl (untransfused)
  * Cardiac: no active ischemia, left ventricular ejection fraction > 45% by MUGA scan
  * Hepatic: bilirubin < 2.0 mg/dl, ALT < 3x the upper limit of normal
  * Pulmonary: FEV1-Forced Expiratory Volume in One Second AND Forced vital capacity (FVC) >50% predicted and Carbon Monoxide Diffusing Capacity (DLCO) (corrected) > 50% predicted
  * Performance status: Karnofsky performance of > 80%.
* Free of active uncontrolled infection at the time of study entry.
* At time of study enrollment > 4 weeks from prior myelosuppressive chemotherapy; and > 6 weeks from prior nitrosoureas.
* Patients must exercise informed voluntary consent and sign a consent form approved by the University of Minnesota IRB: Human Subjects Committee.

Exclusion Criteria:

* Patients will be ineligible if they have advanced myeloma refractory and unresponsive to salvage chemotherapy regimens.
* Female patients who are pregnant (positive b-HCG) or breastfeeding will be excluded from study entry. In addition fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment, particularly after thalidomide will also be excluded from study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2004-04-20 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Brunstein, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemotherapy and Transplant Treatment
Started | 363
Completed | 363
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 363
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 257
  >=65 years | 106
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166
  Male | 197
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 313
  Unknown or Not Reported | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 35
  White | 304
  More than one race | 1
  Unknown or Not Reported | 20
Region of Enrollment [Number; unit: participants]
  United States | 363

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving a Complete Response
Description: Myeloma Response Definitions - Using International Uniform Response Criteria:
  Stringent Complete Response (sCR)requires, plus CR:
  * Normal free light chain ratio
  * Absence of clonal cells in bone marrow
  Complete Response (CR):
  * Absence of the original monoclonal paraprotein
  * <5% plasma cells in a bone marrow aspirate and also on trephine bone biopsy
  * No increase in size or number of lytic bone lesions
  * Disappearance of soft tissue plasmacytomas.
Time Frame: 100 Days post transplant
Population: 173 participants were not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 190
Participants | 51

2. Primary Outcome: Number of Participants Achieving a Complete Response
Description: as for outcome 1
Time Frame: 6 months post transplant
Population: 54 participants were not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 309
Participants | 99

3. Primary Outcome: Number of Participants Achieving a Complete Response
Description: as for outcome 1
Time Frame: 12 months post transplant
Population: 55 participants were not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 308
Participants | 123

4. Secondary Outcome: Number of Patients With Extended Disease-free Survival
Description: Extended disease free survival will be defined as percentage of patients surviving more than 36 months without relapse or disease progression.
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 363
Participants | 164

5. Secondary Outcome: Number of Participants With Overall Survival
Description: The percentage of people in a study or treatment group who are alive for a certain period of time after they were diagnosed with or treated for a disease, such as cancer. Also called survival rate.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 363
Participants | 349

6. Secondary Outcome: Number of Participants With Overall Survival
Description: as for outcome 5
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 363
Participants | 328

7. Secondary Outcome: Number of Participants With Overall Survival
Description: as for outcome 5
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 363
Participants | 301

8. Secondary Outcome: Count of Participants Experiencing Transplant Related Mortality
Description: In the field of transplantation, toxicity is high and all deaths without previous relapse or progression are usually considered as related to transplantation.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 363
Participants | 3

9. Secondary Outcome: Number of Participants Experiencing Incidence of Relapse
Description: The return of disease after its apparent recovery/cessation.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 363
Participants | 69

10. Secondary Outcome: Number of Participants With Disease Progression
Description: Myeloma Response Definitions - Using International Uniform Response Criteria:
  Progressive Disease (PD)
  For patients not in CR or sCR, progressive disease requires one or more of the following:
  * >25% increase in the level of the serum monoclonal paraprotein, which must also be an absolute increase of at least 0.5 g/dL.
  * >25% increase in 24-hour urine protein electrophoresis, which must also be an absolute increase of at least 200 mg/24 hours.
  * Absolute increase in the difference between involved and uninvolved FLC levels (absolute increase must be >10 mg/dl), only in patients without measurable paraprotein in the serum and urine.
  * >25% increase in plasma cells in a bone marrow aspirate or on trephine biopsy, which must also be an absolute increase of at least 10%.
  * Definite increase in the size of existing bone lesions or soft tissue plasmacytomas.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 363
Participants | 34

11. Secondary Outcome: Time to Progression
Description: Mean number of days among patients progressing
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 34
Days | 159.4 (109.8)

12. Secondary Outcome: Time to Relapse
Description: Mean number of days among patients relapsing
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 69
Days | 182.9 (113.5)

13. Secondary Outcome: Number of Participants With Absolute Neutrophil Recovery
Description: Hematologic recovery is defined by absolute neutrophil count (ANC) >2500/μl and platelets > 100,000/μl
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 363
Participants | 363

14. Secondary Outcome: Time to Attainment of CR
Description: Mean (STD) among patients achieving complete remission (CR)
  Myeloma Response Definitions - Using International Uniform Response Criteria:
  Complete Response (CR):
  * Absence of the original monoclonal paraprotein
  * <5% plasma cells in a bone marrow aspirate and also on trephine bone biopsy
  * No increase in size or number of lytic bone lesions
  * Disappearance of soft tissue plasmacytomas
Time Frame: 12 months post transplant
Population: Data was not available on everyone for this endpoint so could only evaluable for 308 out of 363 patients due to data for participants is not available as the EPIC system was not in place when this study was conducted and participants moved to different clinics we do not have follow-up details.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 308
months | 4.6 (1.5)

15. Secondary Outcome: Time to Attainment of CR+PR
Description: Mean (STD) among patients achieving complete remission (CR) and partial remission (PR)
  Myeloma Response Definitions - Using International Uniform Response Criteria:
  Complete Response (CR):
  * Absence of the original monoclonal paraprotein
  * <5% plasma cells in a bone marrow aspirate and also on trephine bone biopsy
  * No increase in size or number of lytic bone lesions
  * Disappearance of soft tissue plasmacytomas.
  Partial Response (PR):
  * Greater than or equal to 50% reduction in the level of the serum monoclonal paraprotein and/or reduction in 24 hour urinary monoclonal paraprotein either by greater than or equal to 90% or to <200 mg/24 hours in light chain disease.
  * If the only measurable non-bone marrow parameter is FLC, greater than or equal to 50% reduction in the difference between involved and uninvolved FLC levels or a 50% decrease in level
Time Frame: 12 months post transplant
Population: 55 patients were not evaluable Data was not available on everyone for this endpoint so could not evaluate all 363 patients
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 308
months | 4.3 (1.5)

16. Secondary Outcome: Duration of Maintenance Treatment
Time Frame: During study
Population: Data not available for this outcome at our center, maintenance treatment data for participants is not available as the EPIC system was not in place when this study was conducted and participants moved to different clinics so follow-up details were no available.
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 0

17. Secondary Outcome: Dropout Rate From Maintenance Therapy
Time Frame: Post transplant phase
Population: as for outcome 16
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 0

18. Secondary Outcome: Number of Participants With Toxicities
Description: Occurrence of toxicities by first 100 days of transplant
Time Frame: By first 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 363
Participants | 68

19. Secondary Outcome: Number of Participants With Infections
Description: Occurrence of infections in the patients by the first 100 days of transplant
Time Frame: By first 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy and Transplant Treatment
Number analyzed (Participants) | 363
Participants | 68

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Chemotherapy and Transplant Treatment
All-Cause Mortality (participants affected / at risk) | 62/363
Serious Adverse Events (participants affected / at risk) | 2/363
Other Adverse Events (participants affected / at risk) | 194/363
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy and Transplant Treatment (N=363)
M-spike increase (Investigations) | 1 (1)
GI bleeding (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy and Transplant Treatment (N=363)
Acute kidney injury (Renal and urinary disorders) | 4 (4)
Akinesis (Nervous system disorders) | 1 (1)
Edema (Renal and urinary disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Artrial fibrillation (Cardiac disorders) | 8 (8)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood clot (Vascular disorders) | 3 (3)
bowl obstruction (Gastrointestinal disorders) | 5 (5)
Cardiomyopathy (Cardiac disorders) | 2 (2)
Cataract (Eye disorders) | 4 (4)
Chest opacities (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Congestive heart failure (Cardiac disorders) | 1 (1)
Cytopenia (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Elevated troponin (Investigations) | 1 (1)
Emphysema (Skin and subcutaneous tissue disorders) | 1 (1)
Encephalopathy (Hepatobiliary disorders) | 1 (1)
Engraftment syndrome (General disorders) | 5 (5)
Epigastric pain (Gastrointestinal disorders) | 1 (1)
Eye hemorrhage (Eye disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
GI bleed (Gastrointestinal disorders) | 8 (8)
GI toxicity (Gastrointestinal disorders) | 1 (1)
Gout (Immune system disorders) | 3 (3)
Hallucinations (Psychiatric disorders) | 2 (2)
Hearing loss (Ear and labyrinth disorders) | 2 (2)
Heart abnormality (Cardiac disorders) | 1 (2)
Hemorrhage (Vascular disorders) | 1 (1)
Hernia (Injury, poisoning and procedural complications) | 2 (2)
Hypercalcemia (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 2 (2)
Hypothyroidism (Investigations) | 1 (1)
Infection (Infections and infestations) | 140 (246)
Intubation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Left hio hemiarhroplasty (Surgical and medical procedures) | 1 (1)
Left vertricular hypertrophy (Cardiac disorders) | 1 (1)
Liver parenchymal disease (Hepatobiliary disorders) | 1 (1)
Low Ejection fraction (Cardiac disorders) | 2 (2)
Macular degeneration (Eye disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 7 (8)
Muscle tear (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 15 (15)
Neurotoxicity (Nervous system disorders) | 3 (3)
Ocular muscle fatigue (Eye disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 4 (4)
Physical Deconditioning (Musculoskeletal and connective tissue disorders) | 3 (3)
Plueral effusions (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 54 (77)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rashes (Skin and subcutaneous tissue disorders) | 1 (1)
Renal calculus (Renal and urinary disorders) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
skin; stevens Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
stent placement for occlusion (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 9 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombosis (Blood and lymphatic system disorders) | 12 (12)
Transminitis (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT00177047/Prot_SAP_000.pdf